CLINICAL TRIAL: NCT02842931
Title: Multicenter, Randomized, Controlled (Comparative), Open, Prospective Study Evaluating an Efficacy of R-DA-EPOCH-21, R-mNHL-BFM-90 and (Auto-SCT)in Patients With DLBCL
Brief Title: R-Dose-adjusted (DA) - EPOCH-21 Versus R-modified Non-Hodgkin Lymphoma (NHL)-Berlin-Frankfurt-Munster (BFM)-90 Program (mNHL-BFM-90) and Autologous Stem Cells Transplantation (Auto-SCT) in DLBCL With Poor Prognosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Collaborators: National Research Center for Hematology (Unknown)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, MD, PhD, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DLBCL-2015
Record Dates: First submitted 2016-03-11; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL, R-DA-EPOCH-21, R-mNHL-BFM-90, auto-SCT
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- R-DA-EPOCH-21 (Active Comparator): Protocol involves 6 cycles.
  Interventions: Drug: R-DA-EPOCH-21
- R-DA-EPOCH-21 + auto-SCT (Active Comparator): Protocol involves 6 cycles. Patients with complete remission undergo auto-SCT after 6 cycles and patients with partial remission after 6 cycles undergo auto-SCT after 2 cycles of R-DHAP
  Interventions: Drug: R-DA-EPOCH-21 + auto-SCT
- R-mNHL-BFM-90 (Active Comparator): Course A:
  Rituximab 375 mg/m2 IV 0 day, Dexamethasone 10 mg/m2/day IV 1 - 5 days, Methotrexate 1000 mg/m2 12 h IV 1 day, Ifosfamide 800 mg/m2/day 1 h IV 1 - 5 days, Etoposide 100 mg/m2/day IV 4, 5 days, Doxorubicin 25 mg/m2/day IV 1, 2 days, Vincristine 2 mg IV 1 day, Cytarabine 100 mg/m2/day IV 1 h 4, 5 days.
  Course B:
  Rituximab 375 mg/m2 IV 0 day, Dexamethasone 10 mg/m2/day IV 1 - 5 days, Cyclophosphamide 200 mg/m2/day IV 1 h 1 - 5 days, Methotrexate 1000 mg/m2 12 h IV 1 day, Doxorubicin 25 mg/m2/day IV 4, 5 days, Vincristine 2 mg IV 1 day. Protocol involves 6 cycles : A-B-A-B-A-B. One cycle continues 21 days.
  Interventions: Drug: R-mNHL-BFM-90
- R-mNHL-BFM-90 + auto-SCT (Active Comparator): Protocol involves 6 cycles R-mNHL-BFM-90: A-B-A-B-A-B. Patients with complete remission undergo auto-SCT after 6 cycles and patients with partial remission after 6 cycles undergo auto-SCT after 2 cycles of R-DHAP
  Interventions: Drug: R-mNHL-BFM-90 + auto-SCT

INTERVENTIONS:
Drug: R-DA-EPOCH-21 — R-DA-EPOCH-21 treatment without auto-SCT for DLBCL patients younger than 60 years with intermediate and high risk for IPI
  Arms: R-DA-EPOCH-21
Drug: R-DA-EPOCH-21 + auto-SCT — R-DA-EPOCH-21 treatment with auto-SCT for DLBCL patients younger than 60 years with intermediate and high risk for IPI
  Arms: R-DA-EPOCH-21 + auto-SCT
Drug: R-mNHL-BFM-90 — R-mNHL-BFM-90 without auto-SCT in patients with DLBCL under the age of 60 years with intermediate and high risk for IPI
  Arms: R-mNHL-BFM-90
Drug: R-mNHL-BFM-90 + auto-SCT — R-mNHL-BFM-90 with auto-SCT in patients with DLBCL under the age of 60 years with intermediate and high risk for IPI
  Arms: R-mNHL-BFM-90 + auto-SCT

SUMMARY:
Purpose: to evaluate an efficacy of chemotherapy regimens R-DA-EPOCH-21 and R-mNHL-BFM-90 with and without autologous hematopoietic stem cells transplantation (auto-SCT) in newly diagnosed patients with DLBCL with intermediate and high risk.

DETAILED DESCRIPTION:
Patients initially are randomized into 4 arms:

1. st arm R-DA-EPOCH-21
2. nd arm R-mNHL-BFM-90
3. rd arm R-DA-EPOCH-21 + auto-SCT
4. th arm of R-mNHL-BFM-90 + auto-SCT

Patients who achieved complete remission after 6 cycles of R-DA-EPOCH-21 or R-mNHL-BFM-90 immunochemotherapy continue to be under observation (1st and 2nd arms) or continue treatment with Rituximab + BCNU+Etoposid+Ara-C+Melphalan (R-BEAM) followed by auto-SCT (3rd and 4th arms). Patients who achieved partial remission after 6 cycles of R-DA-EPOCH-21 or R-mNHL-BFM-90 immunochemotherapy continue treatment with 2 cycles of Rituximab+Dexamethasone+Ara-C+Cisplatin (R-DHAP), continue to be under observation (1st and 2nd arms) or continue treatment with R-BEAM, followed by auto-SCT (3rd and 4th arms).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed DLBCL,
2. No previous treatment with chemotherapy and/or radiation therapy of DLBCL
3. Presence of 2 or more signs of unfavorable prognosis (IPI 2-4)
4. Age 18-60 years.

Exclusion Criteria:

1. Transformation of mature cell lymphomas in DLBCL.
2. B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and Hodgkin's lymphoma
3. B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and Burkitt lymphoma
4. DLBCL of central nervous system (CNS)
5. testicular DLBCL
6. Primary mediastinal large B-cell lymphoma
7. Pretreated DLBCL.
8. HIV-associated DLBCL
9. Congestive heart failure, unstable angina, severe cardiac arrhythmias and conduction disturbances, myocardial infarction.
10. Renal insufficiency (serum creatinine greater than 0.2 mmol/L) (except cases with specific kidney infiltration, urinary tract compression by tumor conglomerate or presence of uric acid nephropathy due to massive cytolysis syndrome).
11. Liver failure (except cases with liver tumor infiltration), acute hepatitis or active phase of chronic hepatitis B or C with serum bilirubin greater than 1.5 standards, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 3 standards, prothrombin index less than 70%.
12. Severe pneumonia (except cases with specific lungs infiltration), accompanied by respiratory failure (dyspnea > 30 in min., hypoxemia less than 70 mm Hg, when it is impossible to compensate situation in 2-3 days).
13. Life-threatening bleeding (gastrointestinal, intracranial), with exception of bleeding due to tumor infiltration of organs (stomach, intestines, uterus, etc.) and disseminated intravascular coagulation due to underlying disease complications after their successful conservative treatment.
14. Severe mental disorders (delusions, severe depressive syndrome and other manifestations of productive symptoms) not related with specific infiltration of central nervous system.
15. Decompensated diabetes.
16. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
complete response | 168 day
  (physical examination, standard blood tests, including assessment of LDH level, thoracic and abdominal computerized tomography (together with any other anatomic site, as clinically indicated), bone marrow biopsy in case of bone marrow involvement and 18F-fludeoxyglucose positron emission tomography (18FDG-PET) (not mandatory) in case of residual measurable disease at the end of the chemoimmunotherapy).

SECONDARY OUTCOMES:
overall survival | Five-year survival
  Survival time and time to disease progression are calculated in months from day of enrollment in the study until death, relapse, progression, or last follow-up, as appropriate
disease-free survival | Five-year survival
  Survival time and time to disease progression are calculated in months from day of enrollment in the study until death, relapse, progression, or last follow-up, as appropriate
event-free survival | Five-year survival
  Survival time and time to disease progression are calculated in months from day of enrollment in the study until death, relapse, progression, or last follow-up, as appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Elena N Parovichnikova, MD PhD, Study Chair — National Research Center for Hematology, Russia
Locations (1):
- National Research Center for Hematology, Moscow, Russia